CLINICAL TRIAL: NCT02925364
Title: Functional and Anatomical MRI of the Spinal Cord and Perispinal Tissues 6 Months After Cardiac Surgery With Standard vs. Gradual Sternal Retraction: Implications for Chronic Post-surgical Pain
Brief Title: Functional and Anatomical MRI of the Spinal Cord and Peri-spinal Tissues
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment
Sponsor: Dr. Tarit Saha (Other)
Responsible Party: Sponsor-Investigator, Dr. Tarit Saha, Director, cardiac anesthesia group, Queen's University
Organization: Queen's University (Other)
Other Study IDs: ANAE-233-13-amendment
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain; Other Functional Disturbances Following Cardiac Surgery
Keywords: magnetic resonance imaging; central pain processing; anatomical MRI; fMRI
MeSH Terms: conditions — Chronic Pain | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No pain: patients who are enrolled in the parent study and report no chest pain at their 6 month post-cardiac surgery follow-up will undergo functional and anatomical MRI
  Interventions: Radiation: magnetic resonance imaging (MRI)
- Pain: Patients who are enrolled in the parent study and report chest pain at their 6 month post-cardiac surgery follow-up will undergo functional and anatomical MRI
  Interventions: Radiation: magnetic resonance imaging (MRI)

INTERVENTIONS:
Radiation: magnetic resonance imaging (MRI) — all participants will undergo a functional MRI and an anatomical MRI in a single session

SUMMARY:
The current study is an amendment to a previously approved blinded randomized controlled trial (NCT02697812) which examines the rate at which the sternal retraction maneuver is performed during cardiac surgery (standard over 30 seconds versus. gradual over 15 minutes) and examines the incidence of chronic post-sternotomy pain 6 months following surgery.

Patients enrolled in the parent study will be identified at the 6 month follow-up and recruited in terms of whether they report chest pain. A total of 30 participants will be recruited (15 with and 15 with no pain) to undergo a single MRI session in which functional MRI will be done on the brain stem and spinal cord and anatomical MRI images will be collected for specific chest and neck structures. This will indicate whether there are long-term differences in pain processing and/or physical damage to neck and chest structures in those with and without chronic pain 6 months following coronary artery bypass graft surgery. All functional and anatomical MRI images will be reviewed and interpreted with study personnel blinded to whether the patient is reporting pain or no pain at their 6 month follow-up interview.

ELIGIBILITY:
Inclusion Criteria:

* Elective Primary Coronary Artery Bypass Surgery
* Understanding and provision of written informed consent
* Age > 18 and < 75
* ASA class I, II or II

Exclusion Criteria:

Any combined or redo cardiac procedure

* Current alcohol or substance abuse
* Pre-existing chronic pain requiring chronic analgesic use
* Rest pain in proposed surgical area at baseline, preoperatively
* Chronic Steroid use
* Inability to perform post-operative assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be those enrolled in a parent blinded randomized controlled trial (NCT02697812). At their 6 month post-cardiac surgery interview, patients reporting no chest pain (n=15) or chest pain (n=15) will be recruited to undergo an MRI.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
functional MRI (fMRI) | 6 months postoperatively
  functional MRI of brain stem & spinal cord

SECONDARY OUTCOMES:
anatomical MRI | 6 months postoperatively
  anatomical MRI of neck & chest

CONTACTS AND LOCATIONS:
Overall Officials: Tarit Saha, MD, FRCPC, Principal Investigator — Queen's University; Patrick Stroman, PhD, Principal Investigator — Queen's University-Cenre for Neuroscience Studies
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No